CLINICAL TRIAL: NCT00227968
Title: Maintenance Therapies in Bipolar Disorder
Brief Title: Psychosocial Therapy Plus Maintenance Pharmacotherapy for Treating Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R37MH029618-95 (NIH); 950310
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Bipolar Disorder
Keywords: Manic-depressive psychosis; Depression, bipolar
MeSH Terms: conditions — Bipolar Disorder

INTERVENTIONS:
Behavioral: Interpersonal Social Rhythm Therapy (IPSRT)
Behavioral: Clinical Status and Symptom Response Therapy (CSSRT)

SUMMARY:
This study will evaluate the effectiveness of interpersonal and social rhythm therapy (IPSRT) versus clinical status and symptom response therapy (CSSRT) in reinforcing the treatment of bipolar disorder in individuals who are currently undergoing medication treatment for the disorder.

DETAILED DESCRIPTION:
Bipolar disorder is a serious medical illness that causes shifts in a person's mood, energy, and ability to function. These changes are drastic, and can result in damaged relationships, poor job or school performance, and suicide. Bipolar disorder is also known as manic-depressive disorder because it is characterized by episodes of mania and depression. Some signs and symptoms of a manic episode include the following: increased energy, activity, and restlessness; excessively "high," overly good mood; and extreme irritability. Some signs and symptoms of a depressive episode include the following: sad, anxious, or empty mood; feelings of hopelessness or pessimism; and feelings of guilt, worthlessness, or helplessness. Bipolar disorder is most effectively treated using a strategy that combines medication and psychosocial treatment. This study will evaluate the effectiveness of IPSRT versus CSSRT in reinforcing the treatment of bipolar disorder in individuals who are currently undergoing maintenance medication treatment for the disorder.

Participants in this open-label study will be randomly assigned to one of two treatment strategies: IPSRT or CSSRT. All participants will attend study visits once a week until they have been stable for 4 weeks (acute phase). At this point, they will attend study visits every other week for 12 weeks (continuation phase), and then once a month for 18 months or until another depressive or mixed episode occurs (maintenance phase). Participants who experience a recurrence will be treated with medication and the type of therapy they were assigned upon study entry (IPSRT or CSSRT). These participants will continue to be followed for a period of time equivalent to their remainder of time in the study had they not experienced a recurrence. Outcomes will be measured at Week 12 of the continuation phase and Week 18 of the maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar disorder
* Currently in the third episode of mania or major depression
* History of one other episode of major depression within 5 years prior to study entry

Exclusion Criteria:

* Currently in the first episode of mania or schizo-affective disorder (manic type)
* Rapid cycling drug or alcohol abuse
* Unstable medical illness
* Pregnant
* Index episode caused by medically prescribed drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181
Dates: Start 1995-03; Study Completion 2002-04

PRIMARY OUTCOMES:
Time to stabilization in the acute phase and time to recurrence in the maintenance phase

SECONDARY OUTCOMES:
Measured at Week 12 of the continuation phase and Week 18 of the maintenance phase: Somatic Symptoms Checklist

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Frank, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Mallinger AG, Frank E, Thase ME, Barwell MM, Diazgranados N, Luckenbaugh DA, Kupfer DJ. Revisiting the effectiveness of standard antidepressants in bipolar disorder: are monoamine oxidase inhibitors superior? Psychopharmacol Bull. 2009;42(2):64-74. PMID 19629023
- [Derived] Frank E, Soreca I, Swartz HA, Fagiolini AM, Mallinger AG, Thase ME, Grochocinski VJ, Houck PR, Kupfer DJ. The role of interpersonal and social rhythm therapy in improving occupational functioning in patients with bipolar I disorder. Am J Psychiatry. 2008 Dec;165(12):1559-65. doi: 10.1176/appi.ajp.2008.07121953. Epub 2008 Oct 1. PMID 18829872